CLINICAL TRIAL: NCT02069093
Title: A Phase II, Single Arm Study of the Use of Steroid-based Mouthwash to Prevent Stomatitis in Postmenopausal Women With Advanced or Metastatic Hormone Receptor Positive Breast Cancer Being Treated With Everolimus Plus Exemestane
Brief Title: Open-label, Phase II Study of Stomatitis Prevention With a Steroid-based Mouthwash in Post-menopausal Women With Estrogen-receptor-positive (ER+), Human Epidermal Growth Factor Receptor 2 (HER2)- Metastatic or Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001JUS226
Record Dates: First submitted 2014-02-20; First posted 2014-02-21 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2016-12

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Everolimus; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexamethasone based mouthwash (Experimental): Participants swished and spat 10mL of 0.5mg/5mL dexamethasone steroid mouthwash (investigational treatment) 4 times daily (qid) orally for 2 minutes each for 8 weeks. Participants remained without food or drink (NPO) for one hour after administration of the mouthwash. Also, participants received everolimus 10 mg and exemstane 25 mg (study treatments) according to local regulations.
  Interventions: Drug: Dexamethasone based mouthwash; Drug: Everolimus; Drug: Exemestane

INTERVENTIONS:
Drug: Dexamethasone based mouthwash — Dexamethasone steroid-based oral solution, comprised of 0.5 milligrams per 5mL of alcohol-free dexamethasone.
Drug: Everolimus — Commercially available everolimus 10 mg was prescribed to participants by the Investigator according to local regulations.
Drug: Exemestane — Commercially available exemestane 25 mg was prescribed to participants by the Investigator according to local regulations.

SUMMARY:
Open-label, Phase II study of Stomatitis prevention with a steroid-based mouthwash in Post-menopausal women with ER+, HER2- Metastatic or Locally Advanced Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Adult women > 18 years of age with metastatic or locally advanced breast cancer not amenable to curative treatment by surgery or radiotherapy
2. Histological or cytological confirmation of hormone-receptor positive (HR+) human epidermal growth factor receptor 2 negative (HER2-) breast cancer
3. Postmenopausal women. Postmenopausal status is defined either by:

   * Age ≥ 55 years and one year or more of amenorrhea
   * Age < 55 years and one year or more of amenorrhea, with an estradiol assay < 20 pg/ml
   * Surgical menopause with bilateral oophorectomy
   * Note: Ovarian radiation or treatment with a luteinizing hormone-releasing hormone (LH-RH) agonist (goserelin acetate or leuprolide acetate) is not permitted for induction of ovarian suppression
4. Patient has been assessed by treating physician to be appropriate candidate for everolimus plus exemestane therapy as treatment of advanced or metastatic breast cancer and plans to prescribe everolimus 10mg PO QD in combination with exemestane 25mg PO QD
5. Patient must start everolimus 10mg plus exemestane 25mg treatment on Cycle 1 Day 1 of trial
6. ECOG Performance status ≤ 2
7. Adequate renal function: serum creatinine ≤ 1.5x ULN;
8. Willingness to self-report level of oral pain using Visual Analog Scale (VAS) and the Normalcy Diet Scale (NDS) throughout each stomatitis event, as required in the patient diary. At baseline, patient's self-reported oral pain level, using VAS, must be 0 and the normalcy diet scale score should ≥ 60
9. Signed informed consent obtained prior to any screening procedure

Exclusion criteria:

1. Patients currently receiving anticancer therapies (except biphosphonate, denosumab);
2. Patients who currently have stomatitis/oral mucositis/mouth ulcers;
3. Known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus);
4. Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral Everolimus;
5. Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary;
6. Patients who have any severe and/or uncontrolled medical conditions such as:

   * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to start of everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
   * Symptomatic congestive heart failure of New York heart Association Class III or IV
   * active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease (except for Hep B and Hep C positive patients)
   * Known severely impaired lung function (spirometry and DLCO 50% or less of normal and O2 saturation 88% or less at rest on room air)
   * active, bleeding diathesis;
7. Chronic treatment with corticosteroids or other immunosuppressive agents. Topical or inhaled corticosteroids are allowed;
8. Known history of HIV seropositivity;
9. Patients who have received live attenuated vaccines within 1 week of start of everolimus and during the study. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines;
10. Patients who have a history of another primary malignancy, with the exceptions of: non-melanoma skin cancer, and carcinoma in situ of the cervix, uteri, or breast from which the patient has been disease free for ≥3 years;
11. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study or patient diaries;
12. Patients who are currently part of any clinical investigation or who has not had resolution of all acute toxic effects or prior anti-cancer therapy to NCI CTCAE version 4.03 Grade 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (23):
  - Highlands Oncology Group Highlands Oncology Group (22), Fayetteville, Arkansas
  - Kaiser Permanente Medical Group Kaiser Permanente-Moanalua M.C, Anaheim, California
  - Los Angeles Hematology/Oncology Medical Group, Los Angeles, California
  - University of California at Los Angeles UCLA and TRIO Network, Los Angeles, California
  - University of California Irvine UC Irvine Medical Center, Orange, California
  - University of California San Francisco UCSF Medical Center, San Francisco, California
  - California Pacific Medical Center SC, San Francisco, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Southeastern Regional Medical Center, Newnan, Georgia
  - OnCare Hawaii, ‘Aiea, Hawaii
  - North Shore University Health System NorthShore University, Evanston, Illinois
  - Oncology Specialists, SC Onc Specialists, Park Ridge, Illinois
  - University of Maryland School of Medicine University of Maryland, Baltimore, Maryland
  - Kaiser Permanente - Mid Atlantic Permanete Research Institut Kaiser Permanente Mid-Atlantic, Rockville, Maryland
  - Karmanos Cancer Institute Karmanos Cancer Institute (2), Detroit, Michigan
  - Saint Luke's Hospital/Marion Bloch Neuroscience Institute Cancer Institute, Kansas City, Missouri
  - Regional Cancer Care Associates Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Hematology Oncology Associates of Northern New Jersey PA DeptofHem-OncofNorthern NJ (2), Morristown, New Jersey
  - M. Francisco Gonzalez, MD.PA Hematology Oncology Center, Columbia, South Carolina
  - Oncology Consultants Oncology Consultants, P.A., Houston, Texas
  - University of Texas/MD Anderson Cancer Center Dept.ofMDAndersonCancerCtr(2), Houston, Texas
  - Delta Oncology Associates Delta Hematology/Oncology, Portsmouth, Virginia
  - Northwest Medical Specialties Northwest Medical - Puyallup, Tacoma, Washington

REFERENCES:
- [Derived] Niikura N, Nakatukasa K, Amemiya T, Watanabe KI, Hata H, Kikawa Y, Taniike N, Yamanaka T, Mitsunaga S, Nakagami K, Adachi M, Kondo N, Shibuya Y, Hayashi N, Naito M, Kashiwabara K, Yamashita T, Umeda M, Mukai H, Ota Y. Oral Care Evaluation to Prevent Oral Mucositis in Estrogen Receptor-Positive Metastatic Breast Cancer Patients Treated with Everolimus (Oral Care-BC): A Randomized Controlled Phase III Trial. Oncologist. 2020 Feb;25(2):e223-e230. doi: 10.1634/theoncologist.2019-0382. Epub 2019 Oct 8. PMID 32043762
- [Derived] Rugo HS, Seneviratne L, Beck JT, Glaspy JA, Peguero JA, Pluard TJ, Dhillon N, Hwang LC, Nangia C, Mayer IA, Meiller TF, Chambers MS, Sweetman RW, Sabo JR, Litton JK. Prevention of everolimus-related stomatitis in women with hormone receptor-positive, HER2-negative metastatic breast cancer using dexamethasone mouthwash (SWISH): a single-arm, phase 2 trial. Lancet Oncol. 2017 May;18(5):654-662. doi: 10.1016/S1470-2045(17)30109-2. Epub 2017 Mar 15. PMID 28314691

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 92 participants were enrolled into the study and received study treatments of everolimus and exemestane. Of these, 86 participants were confirmed to have also received the investigational treatment of dexamethasone steroid mouthwash and comprised the full analysis set (FAS). The patient disposition is based on the FAS.
Period: Overall Study
Arm/Group | Dexamethasone Based Mouthwash
Started | 86
Pharmacokinetic Analysis Set | 50
Completed | 56
Not Completed | 30
Not completed — Disease progression | 14
Not completed — New cancer therapy | 1
Not completed — Death | 1
Not completed — Administrative problems | 1
Not completed — Withdrawal by Subject | 2
Not completed — Abnormal laboratory values | 1
Not completed — Adverse Event | 10

BASELINE CHARACTERISTICS:
Population: Full analysis set: The full analysis set consisted of all participants who received at least one dose of study treatment (everolimus and/or exemestane) and at least one dose of investigational treatment (dexamethasone mouth wash).
Arm/Group | Dexamethasone Based Mouthwash
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.02 (10.921)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stomatitis Grade ≥ 2
Description: The incidence of grade ≥ 2 stomatitis was reported. Grade 1 = minimal symptoms, normal diet; grade 2 = symptomatic, but able to swallow a modified diet; grade 3 = symptomatic and unable to aliment or hydrate orally; and grade 4 = symptoms associated with life-threatening consequences.
Time Frame: 56 days
Population: Full analysis set (FAS): The FAS consisted of all participants who received at least one dose of study treatment (everolimus and/or exemestane) and at least one dose of investigational treatment (dexamethasone mouth wash).
Measure: Number; unit: Participants
Arm/Group | Dexamethasone Based Mouthwash
Number analyzed (Participants) | 86
Participants
  Stomatitis grade >=2: Yes | 2
  Stomatitis grade >=2: No | 83
  Stomatitis grade >=2: Not evaluable | 1
Statistical Analysis 1: Comparison: Dexamethasone Based Mouthwash; A test of the incidence rate R was performed with null hypothesis H0: R>= 0.33 and alternative hypothesis Ha: R<0.33 with a one-sided significance level of 0.05. If the test statistic was negative (actual incidence rate was <0.33), the one-sided p-value for the null hypothesis R>=0.33 was presented. The null hypothesis was rejected if the statistic was negative and the corresponding p-value for the one-sided test was <0.5; Test type: Superiority or Other; p < 0.001, Incidence rate R

2. Secondary Outcome: Time to Resolution of Stomatitis From Grade 2 or Greater to Grade 1 or Less
Description: The number of days to achieve resolution of stomatitis from grade 2 or greater to grade 1 or less was assessed. Grade 1 = minimal symptoms, normal diet; grade 2 = symptomatic, but able to swallow a modified diet; grade 3 = symptomatic and unable to aliment or hydrate orally; and grade 4 = symptoms associated with life-threatening consequences.
Time Frame: 56 days
Population: FAS: The FAS consisted of all participants who received at least one dose of study treatment (everolimus and/or exemestane) and at least one dose of investigational treatment (dexamethasone mouth wash).
Measure: Median (Full Range); unit: Days
Arm/Group | Dexamethasone Based Mouthwash
Number analyzed (Participants) | 86
Days | NA [NA to NA] — Median could not be calculated due to insufficient number of participants with events.

3. Secondary Outcome: Median Number of Mouthwashes Per Day
Description: The median number of mouthwashes per day was assessed.
Time Frame: 56 days
Population: FAS: The FAS set consisted of all participants who received at least one dose of study treatment (everolimus and/or exemestane) and at least one dose of investigational treatment (dexamethasone mouth wash).
Measure: Median (Full Range); unit: Number of mouthwashes
Arm/Group | Dexamethasone Based Mouthwash
Number analyzed (Participants) | 86
Number of mouthwashes | 3.95 [1.9 to 4.0]

4. Secondary Outcome: Number of Participants With All Grades of Stomatitis
Description: The number of participants with all grades of stomatitis was defined as the number of participants who had stomatitis grade 1 or higher. Grade 1 = minimal symptoms, normal diet; grade 2 = symptomatic, but able to swallow a modified diet; grade 3 = symptomatic and unable to aliment or hydrate orally; and grade 4 = symptoms associated with life-threatening consequences.
Time Frame: 56 days
Population: The FAS, consisting of all participants who received at least one dose of study treatment (everolimus and/or exemestane) and at least one dose of investigational treatment (dexamethasone mouth wash), was considered for the analysis. However, only those participants, who were evaluable for stomatitis grade, were analyzed.
Measure: Number; unit: Participants
Arm/Group | Dexamethasone Based Mouthwash
Number analyzed (Participants) | 86
Participants
  Stomatitis all grade | 18
  Not evaluable | 1

5. Secondary Outcome: Dose Intensity of Everolimus and Exemestane
Description: The dose intensity was calculated as the cumulative dose of everolimus or exemestane divided by the length of time on treatment during the first 56 days of treatment.
Time Frame: 56 days
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/day
Arm/Group | Dexamethasone Based Mouthwash
Number analyzed (Participants) | 86
mg/day
  Everolimus | 10.0 [3 to 10]
  Exemestane | 25.0 [8 to 25]

6. Secondary Outcome: Blood Concentration of Everolimus and Exemestane
Description: Blood samples were collected and analyzed.
Time Frame: 28 days (pre-dose)
Population: The PK analysis set, which was a subset of the FAS, was considered for the analysis. However, only participants who had evaluable data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dexamethasone Based Mouthwash
Number analyzed (Participants) | 50
ng/mL
  Everolimus (n=42) | 12.047 (56.492)
  Exemestane (n=48) | 0.657 (234.578)

ADVERSE EVENTS:
Arm/Group | Dexamethasone Based Mouthwash
Serious Adverse Events (participants affected / at risk) | 20/92
Other Adverse Events (participants affected / at risk) | 72/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone Based Mouthwash (N=92)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Generalised oedema (General disorders) | 1
Mass (General disorders) | 1
Pyrexia (General disorders) | 2
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Electrolyte depletion (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Substance abuse (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone Based Mouthwash (N=92)
Anaemia (Blood and lymphatic system disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 14
Oral pain (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 16
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 7
Urinary tract infection (Infections and infestations) | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 14
Hypokalaemia (Metabolism and nutrition disorders) | 5
Dysgeusia (Nervous system disorders) | 12
Headache (Nervous system disorders) | 10
Insomnia (Psychiatric disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.